CLINICAL TRIAL: NCT01777594
Title: A Phase II, Multicenter, Single-Arm Study of G-202 (Mipsagargin) as Second-Line Therapy Following Sorafenib for Adult Patients With Progressive Advanced Hepatocellular Carcinoma
Brief Title: Study of G-202 (Mipsagargin) as Second-Line Therapy Following Sorafenib in Hepatocellular Carcinoma
Acronym: G-202-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GenSpera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-202-003
Record Dates: First submitted 2013-01-18; First posted 2013-01-29 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Advanced Adult Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; HCC; liver; liver cancer; sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G-202 (Mipsagargin) (Experimental): G-202 (mipsagargin) administered by intravenous infusion on 3 consecutive days of a 28-day cycle
  Interventions: Drug: G-202

INTERVENTIONS:
Drug: G-202 — G-202 administered by intravenous infusion (IV, in the vein) on Days 1, 2 and 3 of each 28-day cycle until progression or development of unacceptable toxicity
  Other Names: Mipsagargin

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common type of cancer worldwide and the third most common cause of death from cancer. Sorafenib is the only approved therapy for treatment of advanced HCC, and there is a need to identify more drugs that are beneficial for these patients without unacceptable side effects. Prodrug chemotherapy is an approach in which an inactive non-toxic agent is administered to the patient and gets activated within the body at specific locations, resulting in a higher concentration of the cytotoxic form at a tumor location while avoiding general side effects. G-202 (mipsagargin) is an example of prodrug chemotherapy. It is activated by Prostate Specific Memory Antigen (PSMA), which is expressed by some cancer cells and in the blood vessels of most solid tumors, but not by normal cells or blood vessels in normal tissue. It is believed that activation of the prodrug G-202 will allow the drug to kill cancer cells. This study will evaluate the activity and safety of G-202 in patients with hepatocellular carcinoma who have progressed after taking sorafenib. The study will evaluate clinical activity and safety of G-202 administered by intravenous infusion on three consecutive days of a 28-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent document signed prior to the performance of any study-specific procedures and initiation of study therapy
* At least 18 years of age
* ECOG Performance Status 0 or 1
* Histologic or cytologic confirmation of hepatocellular carcinoma (HCC)
* Child-Pugh score of A or B7
* At least one measurable lesion (preferably in the liver) assessed within 4 weeks of first administration of G-202 by abdominal CT or MRI with dynamic phase imaging of the liver, pelvic CT or MRI with contrast, chest CT with contrast, and bone imaging in patients with known bone metastases or if medically indicated
* Must have received sorafenib therapy and had disease progression on sorafenib therapy or was not able to tolerate sorafenib
* Sorafenib or other anti-cancer therapy must have been discontinued > 21days prior to the first administration of G-202
* Adequate hematologic function (ANC ≥ 1200/mm3, hemoglobin ≥ 8.5 g/dL, platelet count ≥ 75,000/mm3)
* Adequate hepatic function (albumin ≥ 2.8 g/dL, AST and ALT ≤ 5 x ULN, total bilirubin < 2 mg/dL)
* Adequate renal function (proteinuria level ≤ 2+, serum creatinine ≤ 1.5 x ULN)
* Acceptable coagulation profile (PT/INR ≤ 2.3, aPTT ≤ 1.5 x ULN)
* Acute toxicity from previous therapy (excluding alopecia) must have resolved to ≤ Grade 1 per CTCAE v4.0
* Negative serum pregnancy test for women of child-bearing potential

Exclusion Criteria:

* Prior locoregional therapies (e.g., transarterial chemoembolization [TACE]) ≤ 4 weeks prior to the first administration of G-202 or not recovered from treatment-related toxicities.
* Radiotherapy ≤ 4 weeks prior to the first administration of G-202 or not recovered from toxicities (palliative radiotherapy for bone lesions ≤ 2 weeks prior allowed)
* Major surgery ≤ 4 weeks prior to first administration of G-202
* Intolerance to both CT and MRI contrast agents
* Candidate for liver transplantation
* Persistent or untreated biliary infection
* Any GI bleeding within 12 weeks prior to first administration of G-202
* Currently receiving any full-dose anti-coagulation treatment
* Clinically-significant third space fluid accumulation
* Known CNS metastasis, including brain metastasis or leptomeningeal metastasis
* Known human immunodeficiency virus (HIV) positivity
* Viral hepatitis requiring anti-viral therapy
* History or evidence of cardiac risk, including screening QTc interval > 470 msec, clinically-significant uncontrolled arrhythmias or arrhythmia requiring treatment (except atrial fibrillation and paroxysmal supraventricular tachycardia), history of acute coronary syndromes within 6 months (including myocardial infarction and unstable angina, coronary artery bypass graft, angioplasty, or stenting) or history of congestive heart failure with most recent ejection fraction < 45%
* Uncontrolled hypertension (systolic BP ≥ 160 or diastolic BP ≥ 100)
* Cerebrovascular accident or transient ischemic attack within 6 months prior to the first dose of study therapy
* History of pulmonary embolism within 6 months or untreated deep venous thrombosis
* Documentation of keratosis follicularis (also known as Darier or Darier-White disease)
* Requirement for chronic use of inhibitors or inducers of cytochrome (CYP3A4) iso-enzymes
* Known hypersensitivity to any study drug component, including thapsigargin derivatives, polysorbate 20, or propylene glycol
* Known history of another primary malignancy that has not been in remission for at least 2 years (non-melanoma skin cancer, cervical carcinoma in situ or squamous intraepithelial lesions allowed)
* Use of any investigational agent within 4 weeks prior to the first administration of G-202
* Pregnancy or nursing
* Any medical intervention, other medical condition, psychiatric condition or social circumstance which could compromise patient safety and/or adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Time to progression | every 8 weeks, until disease progression (estimated up to 2 years)
  Duration of time from the first administration of G-202 to the time of radiologic progression

SECONDARY OUTCOMES:
Overall response rate | every 8 weeks, until disease progression (estimated up to 2 years)
  Percentage of patients with complete response (CR), partial response (PR) or stable disease (SD) after treatment with G-202
Progression-free survival | every 8-12 weeks, until disease progression or death (estimated up to 3 years)
  Duration of time from the first administration of G-202 to the time of radiologic progression or death
Overall survival | every 12 weeks for approximately 3 years or until patient death
  Duration of time from the first administration of G-202 to the time of death

CONTACTS AND LOCATIONS:
Overall Officials: Devalingam Mahalingam, M.D., Ph.D., Study Chair — University of Texas, Health Science Center, Cancer Therapy and Research Center
Locations (4):
- United States (4):
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Oncology Consultants, PA, Houston, Texas
  - University of Texas Health Sciences Center at Houston, Memorial Hermann Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No